CLINICAL TRIAL: NCT07099339
Title: Effect of Pudendal Nerve Electrical Stimulation on Fecal Incontinence in Children With Repaired Anorectal Malformation: A Randomized Controlled Clinical Trial
Brief Title: Effect of Pudendal Nerve Electrical Stimulation on Fecal Incontinence in Children With Repaired Anorectal Malformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Collaborators: National Institute of Diabetes and Endocrinology, Egypt (Unknown); El Galaa Teaching Hospital (Other); Benha Children Hospital (Other); Benha University (Other)
Responsible Party: Principal Investigator, Amany Gomaa Atiaa, lecturer, Sinai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HB000145
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Fecal Incontinence (FI); Anorectal Malformations
Keywords: Pudendal Nerve Electrical Stimulation; Fecal Incontinence; Children; Repaired; Anorectal Malformation
MeSH Terms: conditions — Fecal Incontinence; Anorectal Malformations | interventions — Behavior Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: the assessor didn't know the grouping of children, intervention received, the data of first assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Control Group children treated by Behavioral Therapy and Kegel Exercise, evaluated by assessing Anal Sphincter Muscle Activity Peak by anal pressure sensor and tracking Defecation Frequency and Fecal Leakage Episodes from the bowel diary.
  Interventions: Behavioral: Behavioral Therapy; Other: Kegel Exercise; Diagnostic Test: Anal Sphincter Muscle Activity Peak; Diagnostic Test: Bowel Diary Documentation
- Study Group (Experimental): Study Group children treated by Behavioral Therapy, Kegel Exercise, and Pudendal Nerve Electrical Stimulation, evaluated by assessing Anal Sphincter Muscle Activity Peak by anal pressure sensor and tracking Defecation Frequency and Fecal Leakage Episodes from the bowel diary.
  Interventions: Behavioral: Behavioral Therapy; Other: Kegel Exercise; Device: Pudendal Nerve Electrical Stimulation; Diagnostic Test: Anal Sphincter Muscle Activity Peak; Diagnostic Test: Bowel Diary Documentation

INTERVENTIONS:
Behavioral: Behavioral Therapy — Behavioral Therapy in form of: Learning and advices, Dietary modifications, Toilet pattern modification, Motivational rewarding system, and Diary documentation.
  Other Names: Cognitive-Behavioral Therapy; Behavioral Modifications
Other: Kegel Exercise — Kegel Exercise done by contracting and relaxing pelvic floor muscles for seconds with hold and repetitions.
  Other Names: Pelvic Floor Muscles Training
Device: Pudendal Nerve Electrical Stimulation — Pudendal Nerve Electrical Stimulation applied bilateral to the right and left pudendal by inserting rectal stimulator electrode anally with the other surface electrode at sacral region.
  Other Names: Anal Electrical Stimulation; Anorectal Electrical Stimulation; Intra-anal Electrical Stimulation
  Arms: Study Group
Diagnostic Test: Anal Sphincter Muscle Activity Peak — Anal Sphincter Muscle Activity Peak was evaluated using anal pressure sensor (in mmHg) = anal squeeze pressure during maximum voluntary contraction - resting anal pressure at rest or resting tone as baseline activity
  Other Names: Pelvic Floor Muscles Activity; Anorectal Manometer
Diagnostic Test: Bowel Diary Documentation — Defecation Frequency and Fecal Leakage Episodes collected from the Bowel Diary that documenting bowel events daily through a period of time "a week".

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effect of pudendal nerve electrical stimulation on fecal incontinence in children with repaired anorectal malformation. Ithe investigators are hypothesized that PNES will significantly improve continence scores, reduce the frequency of fecal incontinent episodes, and enhance the overall quality of life in this vulnerable pediatric population, thereby addressing a critical unmet need in their long-term care.

Children with repaired anorectal malformation may benefit more from combined pudendal nerve electrical stimulation with behavioral therapy and pelvic floor muscles training in improving fecal incontinence.

DETAILED DESCRIPTION:
Anorectal malformation (ARM), commonly known as imperforate anus, represent a spectrum of congenital anomalies where the anus and rectum do not form properly during fetal development, these malformations vary widely in severity, from a simple membrane covering the anal opening to complex defects cloacal malformations involving abnormal connections (fistulas) to the urinary or genital tracts.

Fecal incontinence in this population can stem from various factors, including impaired anorectal sensation, compromised sphincter function, and abnormal bowel motility, severely impacting a child's quality of life, psychosocial development, and integration into social activities.

Current management strategies for FI in children with repaired ARM typically involve a multi-faceted approach, including dietary modifications, laxatives, enemas, and bowel management programs.

Exercises such as Kegels, where children are taught to contract and relax these muscles, are commonly employed to enhance voluntary control and improve the ability to hold stool.

The pudendal nerve plays a vital role in maintaining fecal continence by innervating the external anal sphincter EAS bilaterally by the somatic fibers of the 2nd, 3rd, and 4th sacral roots through its connections to the sacral reflex arc, contributing to rectal sensation, and coordinating pelvic floor muscle function.

All children treated by Behavioral Therapy and Kegel Exercise, and by Pudendal Nerve Electrical Stimulation for the study group.

Outcome Measures: All children were evaluated before the commencement (pretreatment) and after 3 successive months of treatment (posttreatment). The anal sphincter muscle activity peak was assessed by anal pressure sensor and bowel diary was used for tracking defecation frequency and fecal leakage episodes daily.

ELIGIBILITY:
Inclusion Criteria:

* children ages ranged from 6 to 9 years and complain of involuntary leakage of feces with a history of anorectal surgical repair MRI revealed the degree of muscle development "Fair/Hypoplastic" identifiable but less developed or asymmetrical muscles
* they can do minimal palpable voluntary contraction of anal sphincter muscle
* they were able to follow instructions during the testing and treatment procedures.

Exclusion Criteria:

* with severe hypoplasia or complete agenesis/absence of parts of the sphincter complex "Poor/Barely Identifiable/Absent", evidenced by MRI,
* children with post-colon surgery other than ARM, neurologic/neuropathic disorder, spinal cord lesion, sensory or hearing deficits.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Anal Sphincter Muscles Activity Peak | Baseline and after three months
  Anal Sphincter Muscle Activity Peak was evaluated using anal pressure sensor (in mmHg) = anal squeeze pressure during maximum voluntary contraction - resting anal pressure at rest or resting tone as baseline activity.

SECONDARY OUTCOMES:
Defecation Frequency | Baseline and after three months
  Defecation Frequency collected from the bowel diary that documenting bowel events daily through a period of time "a week".
Fecal Leakage Episodes | Baseline and after three months
  Fecal Leakage Episodes collected from the bowel diary that documenting bowel events daily through a period of time "a week".

CONTACTS AND LOCATIONS:
Overall Officials: GOTHI, Study Chair — National Institute for Teaching Hospitals and Institutes
Locations (1):
- General Organization for Teaching Hospitals and Institutes, Cairo, Cairo Governorate, Egypt